CLINICAL TRIAL: NCT03220724
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of EnvSeq-1 and CH505 M5 gp120 Envs Adjuvanted With GLA-SE in Healthy, HIV-Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of EnvSeq-1 and CH505 M5 gp120 Envs Adjuvanted With GLA-SE in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 115; 12042 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A: Group 1 (Experimental): Participants will receive 20 mcg of CH505TF (admixed with GLA-SE) at Months 0, 2, 4, 8, and 12.
  Interventions: Biological: CH505TF; Biological: GLA-SE adjuvant
- Part A: Group 2 (Experimental): Participants will receive 100 mcg of CH505TF (admixed with GLA-SE) at Months 0, 2, 4, 8, and 12.
  Interventions: Biological: CH505TF; Biological: GLA-SE adjuvant
- Part A: Group 3 (Experimental): Participants will receive 400 mcg of CH505TF (admixed with GLA-SE) at Months 0, 2, 4, 8, and 12.
  Interventions: Biological: CH505TF; Biological: GLA-SE adjuvant
- Part A: Group 4 (Placebo Comparator): Participants will receive placebo at Months 0, 2, 4, 8, and 12.
  Interventions: Biological: Placebo
- Part B: Group 5 (Experimental): Participants will receive CH505TF at Month 0; CH505w53 at Month 2; and CH505w78 at Months 4, and 8. GLA-SE adjuvant is admixed with all the CH505 gp120 proteins.
  Interventions: Biological: CH505TF; Biological: CH505w53; Biological: CH505w78; Biological: GLA-SE adjuvant
- Part B: Group 6 (Experimental): Participants will receive CH505TF at Month 0; CH505TF and CH505w53 at Month 2; CH505TF, CH505w53, and CH505w78 at Month 4; CH505w53 and CH505w78 at Month 8. GLA-SE adjuvant is admixed with all the CH505 gp120 proteins.
  Interventions: Biological: CH505TF; Biological: CH505w53; Biological: CH505w78; Biological: GLA-SE adjuvant
- Part B: Group 7 (Experimental): Participants will receive CH505 M5 (admixed with GLA-SE) at Months 0, 2, 4, and 8.
  Interventions: Biological: CH505 M5; Biological: GLA-SE adjuvant
- Part B: Group 8 (Placebo Comparator): Participants will receive placebo at Months 0, 2, 4, and 8.
  Interventions: Biological: Placebo
- Part C: Group 9 (Experimental): Participants will receive CH505TF at Month 0; CH505w53 at Month 2; and CH505w78 at Months 4.
  Interventions: Biological: CH505TF; Biological: CH505w53; Biological: CH505w78

INTERVENTIONS:
Biological: CH505TF — Administered by intramuscular (IM) injection in the thigh
  Other Names: CH505TF gp120
  Arms: Part A: Group 1; Part A: Group 2; Part A: Group 3; Part B: Group 5; Part B: Group 6; Part C: Group 9
Biological: CH505w53 — Administered by IM injection in the thigh
  Other Names: CH505w53 gp120
  Arms: Part B: Group 5; Part B: Group 6; Part C: Group 9
Biological: CH505w78 — Administered by IM injection in the thigh
  Other Names: CH505w78 gp120
  Arms: Part B: Group 5; Part B: Group 6; Part C: Group 9
Biological: CH505 M5 — Administered by IM injection in the thigh
  Other Names: CH505 M5 gp120
  Arms: Part B: Group 7
Biological: GLA-SE adjuvant — Admixed with all CH505 gp120 proteins
  Arms: Part A: Group 1; Part A: Group 2; Part A: Group 3; Part B: Group 5; Part B: Group 6; Part B: Group 7
Biological: Placebo — Administered by IM injection in the thigh
  Arms: Part A: Group 4; Part B: Group 8

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of EnvSeq-1 and CH505 M5 gp120 Envs adjuvanted with GLA-SE in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity of EnvSeq-1 and CH505 M5 gp120 Envs adjuvanted with GLA-SE in healthy, HIV-uninfected adults. The three individual EnvSeq-1 HIV vaccine Envs used in this study are called CH505TF gp120, CH505w53 gp120, and CH505w78 gp120.

This study will take place in two parts: Part A and Part B. Participants in Part A will be randomly assigned to one of four groups. Participants in each group will receive CH505TF (admixed with GLA-SE) or placebo by intramuscular (IM) injection at Months 0, 2, 4, 8, and 12.

Study researchers will evaluate participant data from Part A of the study prior to enrolling participants into Part B of the study. Researchers will also evaluate data from Part A to determine the dosing for Part B.

Participants in Part B will be randomly assigned to one of four groups. Participants in each group will receive IM injections at Months 0, 2, 4, 8. GLA-SE will be admixed with all the CH505 gp120 vaccines. Part B, Group 5 will follow a sequential approach to EnvSeq-1 vaccine administration with administration of the CH505TF vaccine at Month 0, then CH505w53 at Month 2, and CH505w78 at Months 4, and 8. Part B, Group 6 participants will follow an additive approach to EnvSeq-1 administration with administration of the CH505TF vaccine at Month 0; then the CH505TF and CH505w53 vaccines at Month 2; then the CH505TF, CH505w53 and CH505w78 vaccines at Month 4; then the CH505w53 and CH505w78 vaccines at Month 8. Part B, Group 7 participants will receive CH505 M5 at Months 0, 2, 4, and 8. Part B, Group 8 participants will receive placebo injections at each time point.

Additional study visits will occur through Month 18 for participants in Part A and through Month 14 for participants in Part B. Visits may include physical examinations and clinical assessments; blood, urine, and stool collection; HIV testing; risk reduction counseling; and interviews/questionnaires. Study staff will contact participants for follow-up health monitoring at Month 24 for participants in Part A and at Month 20 for participants in Part B.

Part C will be an open-label study arm using the EnvSeq-1 proteins in sequential administration (CH505TF, CH505w53, and CH505w78 gp120s) at the same dose as in Part B (400 mcg) to allow for in-depth analysis of B cell precursor frequency.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria:

* Age of 18 through 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study, completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit
* Willing to be contacted by phone, text message, or e-mail 6 months after completion of the scheduled clinic visits
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

Laboratory Inclusion Values:

Hemogram/Complete Blood Count (CBC):

* Hemoglobin greater than or equal to 11.5 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry:

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology:

* Negative HIV-1 and -2 blood test: Volunteers must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine:

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status:

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (beta-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 115 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 115 study
* Pregnant or breastfeeding
* Active duty and reserve U.S. military personnel

Vaccines and Other Injections:

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 115 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 115 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA or by the national regulatory authority where the volunteer is enrolling. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 115 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 115 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System:

* Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than 60 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease, current or history
* Adverse events of special interest (AESIs)

  * Volunteers who currently have, or have a history of, any condition that could be considered an AESI for the products administered in this protocol (representative examples are listed in the study protocol)
* Immunodeficiency

Clinically Significant Medical Conditions:

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magda Sobieszczyk, Study Chair — Columbia University; James Kobie, Study Chair — University of Alabama at Birmingham
Locations (8):
- United States (8):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Derived] Wolfe LS, Smedley JG 3rd, Bubna N, Hussain A, Harper R, Mostafa S. Development of a platform-based approach for the clinical production of HIV gp120 envelope glycoprotein vaccine candidates. Vaccine. 2021 Jun 29;39(29):3852-3861. doi: 10.1016/j.vaccine.2021.05.073. Epub 2021 Jun 4. PMID 34099325

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: 20 mcg CH505TF mo(0,2,4,8,12)
- Group 2: Vaccine: 100 mcg CH505TF mo(0,2,4,8,12)
- Group 3: Vaccine: 400 mcg CH505TF mo(0,2,4,8,12)
- Group 4: Placebo: Placebo for CH505TF mo(0,2,4,8,12)
- Group 5: Vaccine; Group 9: Vaccine: 400mcg CH505TF(m0), 400mcg CH505w53(
- Group 6: Vaccine: 400mcg CH505TF(m0), 400mcg CH505TF +
- Group 7: Vaccine: 400mcg CH505 M5(m0,2,4,8)
- Group 8: Placebo: Placebo(m0,2,4,8)
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Placebo | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo | Group 9: Vaccine
Started | 12 | 12 | 12 | 6 | 20 | 20 | 20 | 5 | 10
Month 4.5 Immunogenicity Cohort | 11 | 12 | 12 | 3 | 19 | 20 | 19 | 4 | 9
Completed | 9 | 10 | 11 | 3 | 19 | 20 | 18 | 4 | 10
Not Completed | 3 | 2 | 1 | 3 | 1 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 3 | 1 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Placebo | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo | Group 9: Vaccine | Total
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 20 | 20 | 20 | 5 | 10 | 117
Age, Continuous [Median (Full Range); unit: years] | 32 [20 to 48] | 31 [19 to 49] | 27 [20 to 48] | 28 [19 to 45] | 29 [21 to 43] | 28 [18 to 42] | 28 [22 to 48] | 23 [23 to 32] | 30 [19 to 46] | 28 [18 to 49]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 8
  21 - 30 years | 4 | 5 | 7 | 4 | 12 | 11 | 11 | 4 | 4 | 62
  31 - 40 years | 5 | 4 | 2 | 0 | 6 | 5 | 7 | 1 | 3 | 33
  41 - 50 years | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 1 | 14
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 3 | 7 | 9 | 8 | 2 | 5 | 48
  Male | 7 | 7 | 8 | 3 | 13 | 11 | 12 | 3 | 5 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 3 | 3 | 5 | 2 | 2 | 16
  Not Hispanic or Latino | 12 | 11 | 12 | 6 | 17 | 17 | 15 | 3 | 8 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 0 | 2 | 0 | 2 | 1 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 1 | 1 | 1 | 3 | 0 | 0 | 13
  White | 8 | 8 | 6 | 4 | 17 | 16 | 14 | 4 | 7 | 84
  More than one race | 1 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 12 | 12 | 12 | 6 | 20 | 20 | 20 | 5 | 10 | 117

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants Reporting Local Reactogenicity Signs and Symptoms During the Vaccine Regime
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017], The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through Month Measured through 7 days after the vaccination at Month 0, 2, 4, 8, 12
Measure: Count of Participants; unit: Participants
Groups:
- Part A, Group 1: Vaccine: 20 mcg CH505TF mo(0,2,4,8,12)
- Part A, Group 2: Vaccine: 100 mcg CH505TF mo(0,2,4,8,12)
- Part A, Group 3: Vaccine: 400 mcg CH505TF mo(0,2,4,8,12)
- Part A, Group 4: Placebo: Placebo for CH505TF mo(0,2,4,8,12)
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  Pain: None | 1 | 0 | 2 | 5
  Pain: Mild | 7 | 8 | 6 | 1
  Pain: Moderate | 3 | 4 | 4 | 0
  Pain: Severe | 1 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 1 | 3 | 0 | 6
  Tenderness: Mild | 6 | 5 | 7 | 0
  Tenderness: Moderate | 5 | 4 | 5 | 0
  Tenderness: Severe | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 1 | 0 | 0 | 5
  Pain and/or Tenderness: Mild | 6 | 7 | 7 | 1
  Pain and/or Tenderness: Moderate | 4 | 5 | 5 | 0
  Pain and/or Tenderness: Severe | 1 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema/Redness: None | 10 | 9 | 10 | 5
  Erythema/Redness: Mild | 1 | 2 | 1 | 1
  Erythema/Redness: Moderate | 1 | 0 | 0 | 0
  Erythema/Redness: Severe | 0 | 1 | 1 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Induration/Swelling: None | 11 | 9 | 11 | 6
  Induration/Swelling: Mild | 0 | 0 | 0 | 0
  Induration/Swelling: Moderate | 1 | 2 | 0 | 0
  Induration/Swelling: Severe | 0 | 1 | 1 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 10 | 8 | 10 | 5
  Erythema and/or Induration: Mild | 1 | 1 | 1 | 1
  Erythema and/or Induration: Moderate | 1 | 2 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 1 | 1 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms During the Vaccine Regime
Description: as for outcome 1
Time Frame: Measured through Month Measured through 7 days after the vaccination at Month 0, 2, 4, 8, 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  Malaise and/or fatigue: None | 5 | 4 | 5 | 4
  Malaise and/or fatigue: Mild | 3 | 4 | 5 | 2
  Malaise and/or fatigue: Moderate | 4 | 4 | 2 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 6 | 7 | 9 | 6
  Myalgia: Mild | 4 | 4 | 2 | 0
  Myalgia: Moderate | 2 | 1 | 1 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 8 | 7 | 6 | 5
  Headache: Mild | 2 | 4 | 4 | 1
  Headache: Moderate | 2 | 0 | 1 | 0
  Headache: Severe | 0 | 1 | 1 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 9 | 10 | 11 | 5
  Nausea: Mild | 2 | 2 | 0 | 0
  Nausea: Moderate | 1 | 0 | 1 | 1
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 12 | 12 | 12 | 5
  Vomiting: Mild | 0 | 0 | 0 | 1
  Vomiting: Moderate | 0 | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 10 | 11 | 11 | 5
  Chills: Mild | 1 | 1 | 1 | 1
  Chills: Moderate | 1 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 7 | 8 | 10 | 5
  Arthralgia: Mild | 4 | 3 | 1 | 1
  Arthralgia: Moderate | 1 | 1 | 1 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 4 | 2 | 3 | 3
  Max. Systemic Symptoms: Mild | 4 | 5 | 5 | 2
  Max. Systemic Symptoms: Moderate | 4 | 4 | 3 | 1
  Max. Systemic Symptoms: Severe | 0 | 1 | 1 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Temperature: None | 12 | 10 | 11 | 6
  Temperature: Mild | 0 | 1 | 1 | 0
  Temperature: Moderate | 0 | 1 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity During the Vaccine Regime
Description: From the study termination form, early termination reasons associated with an AE or reactogenicity are tabulated by treatment arm
Time Frame: Measured through Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through the Month 12 boost
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  Clinical Event | 1 | 1 | 0 | 0
  Reactogenicity | 0 | 0 | 0 | 0
  Other reason | 2 | 2 | 1 | 2
  No discontinuation | 9 | 9 | 11 | 4

5. Primary Outcome: Part A: Chemistry and Hematology Laboratory Measures, for Each Boost: Alkaline Phosphatase, AST, ALT in U/L
Description: Laboratory results are summarized by analyte and timepoint. Analytes and timepoint combinations with no grade 1 or higher results are not shown.
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, 8, 12, and at Month 15
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
U/L
  ALT (SGPT) (U/L)- Screening | 18.5 [13 to 24.5] | 20.5 [18 to 24.5] | 22 [17 to 27.5] | 19 [15 to 21]
  ALT (SGPT) (U/L)- Day 14: number analyzed (Participants) | 12 | 12 | 12 | 5
  ALT (SGPT) (U/L)- Day 14 | 19 [13 to 25.5] | 18 [12.5 to 23.5] | 19.5 [17 to 21.5] | 15 [14 to 24]
  ALT (SGPT) (U/L)- Day 70: number analyzed (Participants) | 11 | 12 | 12 | 3
  ALT (SGPT) (U/L)- Day 70 | 19 [13 to 26] | 18 [13.5 to 24.5] | 16.5 [15.5 to 27.5] | 18 [9 to 18]
  ALT (SGPT) (U/L)- Day 126: number analyzed (Participants) | 11 | 12 | 12 | 3
  ALT (SGPT) (U/L)- Day 126 | 18 [15 to 23] | 16 [11 to 25] | 18.5 [14.5 to 23] | 15 [14 to 24]
  ALT (SGPT) (U/L)- Day 238: number analyzed (Participants) | 11 | 11 | 10 | 4
  ALT (SGPT) (U/L)- Day 238 | 16 [13 to 23] | 14 [11 to 25] | 18 [16 to 21] | 16.5 [13.5 to 23.5]
  ALT (SGPT) (U/L)- Day 378: number analyzed (Participants) | 9 | 11 | 11 | 4
  ALT (SGPT) (U/L)- Day 378 | 16 [15 to 19] | 15 [13 to 30] | 18 [16 to 41] | 21.5 [16 to 43]
  ALT (SGPT) (U/L)- Day 455: number analyzed (Participants) | 10 | 11 | 11 | 4
  ALT (SGPT) (U/L)- Day 455 | 20.5 [12 to 30] | 27 [15 to 36] | 14 [13 to 24] | 22.5 [14 to 38]
  AST (U/L)- Screening | 24.5 [18.5 to 35.5] | 22.5 [19 to 27.5] | 22.5 [18.5 to 27.5] | 20 [16 to 27]
  AST (U/L)- Day 14: number analyzed (Participants) | 12 | 12 | 12 | 5
  AST (U/L)- Day 14 | 23.5 [19 to 27] | 22 [18.5 to 24.5] | 22 [19 to 23.5] | 22 [14 to 24]
  AST (U/L)- Day 70: number analyzed (Participants) | 11 | 12 | 12 | 3
  AST (U/L)- Day 70 | 22 [19 to 27] | 21.5 [18 to 24] | 20.5 [18.5 to 25] | 17 [15 to 27]
  AST (U/L)- Day 126: number analyzed (Participants) | 11 | 12 | 12 | 3
  AST (U/L)- Day 126 | 20 [19 to 25] | 20.5 [15.5 to 24] | 19 [15 to 23.5] | 23 [15 to 30]
  AST (U/L)- Day 238: number analyzed (Participants) | 11 | 11 | 10 | 4
  AST (U/L)- Day 238 | 22 [19 to 25] | 20 [16 to 26] | 20 [19 to 24] | 21 [18.5 to 27]
  AST (U/L)- Day 378: number analyzed (Participants) | 9 | 11 | 11 | 4
  AST (U/L)- Day 378 | 22 [17 to 27] | 20 [16 to 26] | 23 [16 to 28] | 22 [17.5 to 45]
  AST (U/L)- Day 455: number analyzed (Participants) | 10 | 11 | 11 | 4
  AST (U/L)- Day 455 | 20 [17 to 33] | 26 [22 to 35] | 20 [16 to 24] | 24 [18.5 to 32]
  Alkaline Phosphatase (U/L)- Screening | 64.5 [52 to 71.5] | 62.5 [55.5 to 81] | 63 [51 to 67] | 66.5 [55 to 81]
  Alkaline Phosphatase (U/L)- Day 14: number analyzed (Participants) | 12 | 12 | 12 | 5
  Alkaline Phosphatase (U/L)- Day 14 | 61.5 [51.5 to 68] | 58.5 [55.5 to 79] | 68.5 [52 to 75] | 58 [55 to 66]
  Alkaline Phosphatase (U/L)- Day 70: number analyzed (Participants) | 11 | 12 | 12 | 3
  Alkaline Phosphatase (U/L)- Day 70 | 60 [48 to 70] | 61.5 [52 to 79] | 64.5 [56 to 73.5] | 67 [54 to 112]
  Alkaline Phosphatase (U/L)- Day 126: number analyzed (Participants) | 11 | 12 | 12 | 3
  Alkaline Phosphatase (U/L)- Day 126 | 65 [49 to 74] | 65 [52.5 to 77.5] | 64.5 [55.5 to 77] | 69 [45 to 71]
  Alkaline Phosphatase (U/L)- Day 238: number analyzed (Participants) | 11 | 11 | 10 | 4
  Alkaline Phosphatase (U/L)- Day 238 | 66 [50 to 79] | 61 [55 to 77] | 67 [57 to 78] | 57 [47.5 to 68]
  Alkaline Phosphatase (U/L)- Day 378: number analyzed (Participants) | 9 | 11 | 11 | 4
  Alkaline Phosphatase (U/L)- Day 378 | 69 [61 to 71] | 74 [56 to 89] | 66 [63 to 75] | 61.5 [55.5 to 68]
  Alkaline Phosphatase (U/L)- Day 455: number analyzed (Participants) | 10 | 11 | 11 | 4
  Alkaline Phosphatase (U/L)- Day 455 | 61.5 [59 to 82] | 67 [59 to 75] | 63 [56 to 73] | 62 [53.5 to 75.5]

6. Primary Outcome: Part A: Chemistry and Hematology Laboratory Measures, for Each Boost: Hemoglobin, Creatinine in g/dL
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, 8, 12, and at Month 15
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
g/dL
  Hemoglobin (g/dL)- Screening | 14 [13.55 to 14.9] | 14.5 [13.75 to 15.3] | 14.6 [13.3 to 15.8] | 13.75 [12.6 to 15.4]
  Hemoglobin (g/dL)- Day 14: number analyzed (Participants) | 12 | 12 | 12 | 5
  Hemoglobin (g/dL)- Day 14 | 13.6 [13 to 14.7] | 13.6 [12.8 to 14.95] | 14.15 [13 to 15.4] | 12.3 [11.8 to 15.1]
  Hemoglobin (g/dL)- Day 70: number analyzed (Participants) | 11 | 12 | 12 | 3
  Hemoglobin (g/dL)- Day 70 | 14 [13.4 to 15.3] | 14.35 [12.45 to 14.8] | 14.65 [12.95 to 15.7] | 12.7 [11 to 15.6]
  Hemoglobin (g/dL)- Day 126: number analyzed (Participants) | 11 | 12 | 12 | 3
  Hemoglobin (g/dL)- Day 126 | 13.7 [13.4 to 15.4] | 14.25 [12.55 to 14.95] | 14.7 [12.5 to 15.25] | 12.7 [11.6 to 13.1]
  Hemoglobin (g/dL)- Day 238: number analyzed (Participants) | 11 | 10 | 10 | 4
  Hemoglobin (g/dL)- Day 238 | 13.8 [13.3 to 14.6] | 14.2 [13.2 to 14.9] | 14.9 [14.2 to 15.3] | 11.75 [11.1 to 13.75]
  Hemoglobin (g/dL)- Day 378: number analyzed (Participants) | 9 | 11 | 11 | 4
  Hemoglobin (g/dL)- Day 378 | 13.8 [13.7 to 15] | 14.3 [12.3 to 14.8] | 14.4 [13.9 to 15.6] | 12.2 [11.1 to 14.4]
  Hemoglobin (g/dL)- Day 455: number analyzed (Participants) | 10 | 11 | 11 | 4
  Hemoglobin (g/dL)- Day 455 | 13.8 [13.6 to 15] | 13.8 [12.9 to 15.1] | 14.5 [13.4 to 15.4] | 12.45 [12 to 13.45]
  Creatinine (g/dL)- Screening | 0.000885 [0.000775 to 0.00102] | 0.00094 [0.000725 to 0.001075] | 0.000905 [0.000785 to 0.000985] | 0.00082 [0.00069 to 0.0011]
  Creatinine (g/dL)- Day 14: number analyzed (Participants) | 11 | 12 | 12 | 5
  Creatinine (g/dL)- Day 14 | 0.00081 [0.0008 to 0.001] | 0.000935 [0.00078 to 0.001145] | 0.0009 [0.000845 to 0.00101] | 0.00072 [0.00066 to 0.00092]
  Creatinine (g/dL)- Day 70: number analyzed (Participants) | 11 | 11 | 12 | 3
  Creatinine (g/dL)- Day 70 | 0.0009 [0.00078 to 0.00097] | 0.00087 [0.0008 to 0.00111] | 0.000905 [0.0008 to 0.000965] | 0.00083 [0.00054 to 0.0011]
  Creatinine (g/dL)- Day 126: number analyzed (Participants) | 11 | 12 | 12 | 3
  Creatinine (g/dL)- Day 126 | 0.00088 [0.0008 to 0.00102] | 0.00102 [0.0008 to 0.00109] | 0.0009 [0.00087 to 0.001] | 0.00081 [0.00061 to 0.00086]
  Creatinine (g/dL)- Day 238: number analyzed (Participants) | 11 | 11 | 9 | 4
  Creatinine (g/dL)- Day 238 | 0.00084 [0.00072 to 0.00104] | 0.00089 [0.00076 to 0.00109] | 0.00084 [0.00082 to 0.0009] | 0.00072 [0.00067 to 0.00084]
  Creatinine (g/dL)- Day 378: number analyzed (Participants) | 9 | 11 | 11 | 4
  Creatinine (g/dL)- Day 378 | 0.00085 [0.0008 to 0.00094] | 0.0009 [0.0008 to 0.00109] | 0.0009 [0.00077 to 0.001] | 0.000695 [0.000615 to 0.00086]
  Creatinine (g/dL)- Day 455: number analyzed (Participants) | 10 | 11 | 11 | 4
  Creatinine (g/dL)- Day 455 | 0.0008 [0.00076 to 0.00094] | 0.00101 [0.00076 to 0.00105] | 0.0009 [0.0008 to 0.00098] | 0.000675 [0.00064 to 0.000795]

7. Primary Outcome: Part A: Chemistry and Hematology Laboratory Measures, for Each Boost: WBC, Platelets, Lymphocytes, Neutrophils
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, 8, 12, and at Month 15
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: 1000 cells per mm^3
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
1000 cells per mm^3
  Platelets (1000 cells per mm^3)- Screening | 226.5 [196 to 270] | 229.95 [206.7 to 258] | 249.35 [229.5 to 282] | 262.8 [230.5 to 300]
  Platelets (1000 cells per mm^3)- Day 14: number analyzed (Participants) | 12 | 12 | 12 | 5
  Platelets (1000 cells per mm^3)- Day 14 | 243 [192 to 265.75] | 232.85 [218.5 to 269.65] | 264.5 [245.5 to 302.9] | 289 [273 to 292]
  Platelets (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 11 | 12 | 12 | 3
  Platelets (1000 cells per mm^3)- Day 70 | 231 [215.4 to 263.2] | 222 [210.5 to 251] | 265.5 [241.05 to 294] | 336 [235.6 to 351]
  Platelets (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 11 | 12 | 12 | 2
  Platelets (1000 cells per mm^3)- Day 126 | 251 [214 to 273] | 218 [208.95 to 276] | 252.5 [235.5 to 275.35] | 326.5 [296 to 357]
  Platelets (1000 cells per mm^3)- Day 238: number analyzed (Participants) | 11 | 10 | 10 | 4
  Platelets (1000 cells per mm^3)- Day 238 | 250 [199 to 262] | 224.5 [217 to 287] | 252.5 [239.6 to 270] | 295.5 [223.5 to 329.5]
  Platelets (1000 cells per mm^3)- Day 378: number analyzed (Participants) | 9 | 11 | 11 | 4
  Platelets (1000 cells per mm^3)- Day 378 | 252 [215.1 to 266] | 230 [203 to 273] | 247 [213 to 278.9] | 293.5 [224.5 to 314.5]
  Platelets (1000 cells per mm^3)- Day 455: number analyzed (Participants) | 10 | 11 | 11 | 4
  Platelets (1000 cells per mm^3)- Day 455 | 236 [222 to 248] | 219 [204 to 247] | 245.4 [225 to 301] | 294 [231 to 327]

8. Primary Outcome: Part A: Occurrence of HIV-specific IgG Responses 2 Weeks After the Third Vaccination With CH505TF gp120
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation.
Time Frame: Measured at Month 4.5
Population: "Overall Number of Participants Analyzed" includes the HIV uninfected participants with samples collected at the month 4.5 immunogenicity timepoint. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  1086C_D7gp120.avi/293F at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  1086C_D7gp120.avi/293F at Month 4.5 | 8 | 8 | 9 | 0
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5 | 8 | 8 | 9 | 0
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5 | 8 | 8 | 9 | 0
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5 | 8 | 8 | 9 | 0
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5 | 8 | 8 | 9 | 0
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  Con 6 gp120/B at Month 4.5 | 8 | 8 | 9 | 0
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  Con S gp140 CFI at Month 4.5 | 8 | 8 | 8 | 0
  gp41 at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  gp41 at Month 4.5 | 0 | 0 | 0 | 0

9. Primary Outcome: Part A: Level of HIV-specific IgG Responses 2 Weeks After the Third Vaccination With CH505TF gp120
Description: as for outcome 8
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
relative fluorescence units
  1086C_D7gp120.avi/293F at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  1086C_D7gp120.avi/293F at Month 4.5 | 27266.375 [24133.25 to 29136.875] | 27854.25 [22628 to 28870.5] | 28419.25 [28098.25 to 29462.25] | 1 [1 to 4.25]
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5 | 24789.25 [18116.75 to 27759.25] | 26439.75 [7317.75 to 27026.25] | 26973 [25791.25 to 27904.5] | 1 [1 to 23.25]
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5 | 15775.25 [6227.25 to 26555] | 17409.5 [1869.5 to 22388.75] | 22807.5 [17251 to 24569.5] | 1 [1 to 15]
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5 | 10859.875 [1526.375 to 24698.625] | 7335.75 [336.25 to 8839] | 10491.75 [6053.5 to 18757.25] | 1 [1 to 19]
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5 | 21460.5 [13024.375 to 27776.375] | 24931 [4200.75 to 26381.75] | 25146 [24498 to 27011] | 1 [1 to 11.5]
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  Con 6 gp120/B at Month 4.5 | 11897.375 [782.875 to 25171.625] | 3169.25 [297 to 15782] | 14748.5 [4326 to 21312.25] | 1 [1 to 1]
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  Con S gp140 CFI at Month 4.5 | 5229.75 [1455.375 to 26839.375] | 12523.25 [400.5 to 19679.75] | 15397 [6772.25 to 24537.25] | 1 [1 to 1]
  gp41 at Month 4.5: number analyzed (Participants) | 8 | 9 | 9 | 3
  gp41 at Month 4.5 | 1 [1 to 2.375] | 1 [1 to 20.25] | 72.5 [1 to 208] | 92.5 [1 to 2345.75]

10. Primary Outcome: Part A: Occurrence of HIV-specific IgA Responses 2 Weeks After the Third Vaccination With CH505TF gp120
Description: Serum HIV-1-specific IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation.
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  1086C_D7gp120.avi/293F at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  1086C_D7gp120.avi/293F at Month 4.5 | 8 | 6 | 11 | 0
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5 | 8 | 6 | 9 | 0
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5 | 8 | 4 | 8 | 0
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5 | 5 | 3 | 5 | 0
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5 | 8 | 6 | 9 | 0
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  Con 6 gp120/B at Month 4.5 | 3 | 2 | 4 | 0
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  Con S gp140 CFI at Month 4.5 | 4 | 3 | 4 | 0
  gp41 at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  gp41 at Month 4.5 | 0 | 0 | 0 | 0

11. Primary Outcome: Part A: Level of HIV-specific IgA Responses 2 Weeks After the Third Vaccination With CH505TF gp120
Description: as for outcome 10
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
relative fluorescence units
  1086C_D7gp120.avi/293F at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  1086C_D7gp120.avi/293F at Month 4.5 | 1379.5 [114.25 to 7947.5] | 3116.125 [528.75 to 8968.125] | 3498 [2746.25 to 4777] | 1 [1 to 1]
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH0505_CON D7gp120_D368R_avi/293F/Mon at Month 4.5 | 1812 [315 to 4170.25] | 1718.5 [135.875 to 3705.375] | 2684.5 [1163.75 to 5112.25] | 1 [1 to 100.5]
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH0505_CON D7gp120_avi/293F/Mon at Month 4.5 | 684.375 [162.25 to 1813] | 658.625 [47 to 1495.5] | 985 [384.5 to 1225.75] | 1 [1 to 196.5]
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH505TF D7gp120d371_avi/293F/Mon at Month 4.5 | 174.625 [1 to 490.25] | 89.125 [10.875 to 858] | 109.25 [1 to 503.5] | 1 [1 to 261.75]
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  CH505TFD8N156KN160K_avi/293i Mon at Month 4.5 | 1142.5 [256.25 to 2757] | 1065.875 [78.375 to 2239.25] | 1594 [689.75 to 1869.25] | 1 [1 to 182]
  Con 6 gp120/B at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  Con 6 gp120/B at Month 4.5 | 18.25 [1 to 164.75] | 26.25 [1 to 196.125] | 75.25 [1 to 621.75] | 1 [1 to 16.75]
  Con S gp140 CFI at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  Con S gp140 CFI at Month 4.5 | 14.25 [1 to 347.75] | 28.875 [1 to 1597.875] | 3 [1 to 347.75] | 1 [1 to 1]
  gp41 at Month 4.5: number analyzed (Participants) | 10 | 8 | 11 | 3
  gp41 at Month 4.5 | 1 [1 to 8.75] | 1 [1 to 26.375] | 1 [1 to 21.25] | 1 [1 to 264.75]

12. Primary Outcome: Number of Part B Participants Reporting Local Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through Month Measured through Month Measured through 7 days after the vaccination at Month 0, 2, 4, 8
Measure: Count of Participants; unit: Participants
Groups:
- Group 5: Vaccine: 400mcg CH505TF(m0), 400mcg CH505w53(m2), 400mcg CH505w78(m4,8)
- Group 6: Vaccine: 400mcg CH505TF(m0), 400mcg CH505TF + CH505W53(m2), 400mcg CH505TF + CH505w53 + CH505w78(m4), 400mcg CH505w53 + CH505w78(m8)
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
Participants
  Pain: None | 4 | 3 | 0 | 4
  Pain: Mild | 9 | 12 | 14 | 1
  Pain: Moderate | 5 | 5 | 4 | 0
  Pain: Severe | 2 | 0 | 2 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 2 | 0 | 0 | 3
  Tenderness: Mild | 11 | 17 | 14 | 2
  Tenderness: Moderate | 6 | 2 | 5 | 0
  Tenderness: Severe | 1 | 1 | 1 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 2 | 0 | 0 | 3
  Pain and/or Tenderness: Mild | 10 | 13 | 13 | 2
  Pain and/or Tenderness: Moderate | 6 | 6 | 5 | 0
  Pain and/or Tenderness: Severe | 2 | 1 | 2 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema/Redness: None | 15 | 16 | 13 | 5
  Erythema/Redness: Mild | 1 | 3 | 2 | 0
  Erythema/Redness: Moderate | 2 | 1 | 3 | 0
  Erythema/Redness: Severe | 2 | 0 | 2 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Induration/Swelling: None | 14 | 15 | 14 | 5
  Induration/Swelling: Mild | 1 | 2 | 1 | 0
  Induration/Swelling: Moderate | 4 | 2 | 3 | 0
  Induration/Swelling: Severe | 1 | 1 | 2 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 14 | 15 | 12 | 5
  Erythema and/or Induration: Mild | 1 | 2 | 3 | 0
  Erythema and/or Induration: Moderate | 3 | 2 | 2 | 0
  Erythema and/or Induration: Severe | 2 | 1 | 3 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Part B Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through Month Measured through Month Measured through 7 days after the vaccination at Month 0, 2, 4, 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
Participants
  Malaise and/or fatigue: None | 7 | 5 | 3 | 3
  Malaise and/or fatigue: Mild | 4 | 9 | 12 | 2
  Malaise and/or fatigue: Moderate | 6 | 5 | 4 | 0
  Malaise and/or fatigue: Severe | 3 | 1 | 1 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 11 | 8 | 6 | 4
  Myalgia: Mild | 1 | 8 | 9 | 0
  Myalgia: Moderate | 7 | 4 | 5 | 1
  Myalgia: Severe | 1 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 8 | 9 | 6 | 2
  Headache: Mild | 8 | 9 | 8 | 3
  Headache: Moderate | 3 | 2 | 6 | 0
  Headache: Severe | 1 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 12 | 15 | 14 | 4
  Nausea: Mild | 7 | 4 | 5 | 1
  Nausea: Moderate | 1 | 1 | 1 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 19 | 20 | 20 | 5
  Vomiting: Mild | 0 | 0 | 0 | 0
  Vomiting: Moderate | 1 | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 12 | 14 | 12 | 5
  Chills: Mild | 5 | 6 | 6 | 0
  Chills: Moderate | 2 | 0 | 2 | 0
  Chills: Severe | 1 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 12 | 17 | 15 | 5
  Arthralgia: Mild | 5 | 3 | 4 | 0
  Arthralgia: Moderate | 2 | 0 | 1 | 0
  Arthralgia: Severe | 1 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 5 | 1 | 1 | 1
  Max. Systemic Symptoms: Mild | 4 | 11 | 11 | 3
  Max. Systemic Symptoms: Moderate | 8 | 7 | 7 | 1
  Max. Systemic Symptoms: Severe | 3 | 1 | 1 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Temperature: None | 17 | 19 | 18 | 5
  Temperature: Mild | 2 | 1 | 2 | 0
  Temperature: Moderate | 1 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0

14. Primary Outcome: Part B: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity During the Vaccine Regime
Description: as for outcome 3
Time Frame: Measured through Month 20
Measure: Count of Participants; unit: Participants
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
Participants | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Part B Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through the Month 8 boost
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
Participants
  Reactogenicity symptoms | 1 | 0 | 0 | 0
  Withdrawal by Subject | 0 | 0 | 0 | 0
  Investigator reason | 1 | 0 | 0 | 0
  Lost to Follow-Up | 1 | 0 | 0 | 1
  Did not discontinue SPA | 17 | 20 | 20 | 4

16. Primary Outcome: Part B Chemistry and Hematology Laboratory Measures, for Each Boost: Alkaline Phosphatase, AST, ALT in U/L
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, 8, and at Month 11
Population: T5-T8 All enrolled
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
U/L
  ALT (SGPT) (U/L)- Screening | 16 [12.5 to 19.5] | 18.5 [13.5 to 28] | 16.5 [12 to 28] | 16 [14 to 23]
  ALT (SGPT) (U/L)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  ALT (SGPT) (U/L)- Day 14 | 14.5 [12 to 19] | 18 [13 to 21.5] | 17 [12 to 31] | 15 [15 to 17]
  ALT (SGPT) (U/L)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  ALT (SGPT) (U/L)- Day 70 | 13 [12 to 22] | 18 [11 to 24] | 15 [12 to 23] | 18.5 [10.5 to 28]
  ALT (SGPT) (U/L)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  ALT (SGPT) (U/L)- Day 126 | 14 [13 to 17] | 18.5 [13.5 to 28.5] | 17 [13 to 24] | 22 [12 to 30.5]
  ALT (SGPT) (U/L)- Day 238: number analyzed (Participants) | 17 | 18 | 18 | 4
  ALT (SGPT) (U/L)- Day 238 | 16 [12 to 22] | 18.5 [10 to 28] | 14.5 [12 to 30] | 15 [11 to 34]
  ALT (SGPT) (U/L)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  ALT (SGPT) (U/L)- Day 308 | 14.5 [12 to 18] | 20 [13.5 to 26] | 19 [15 to 30] | 14.5 [11 to 31.5]
  AST (U/L)- Screening | 19 [17.5 to 23] | 22 [20 to 23.5] | 18 [16.5 to 29] | 20 [17 to 23]
  AST (U/L)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  AST (U/L)- Day 14 | 18 [15.5 to 24.5] | 21 [17.5 to 23] | 18 [15 to 25] | 18 [17 to 21]
  AST (U/L)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  AST (U/L)- Day 70 | 20 [16 to 22] | 19 [17 to 24] | 18 [16 to 22] | 19 [14.5 to 20]
  AST (U/L)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  AST (U/L)- Day 126 | 18 [16 to 23] | 20.5 [18.5 to 27] | 19 [16 to 24] | 18.5 [14 to 23.5]
  AST (U/L)- Day 238: number analyzed (Participants) | 17 | 18 | 18 | 4
  AST (U/L)- Day 238 | 18 [15 to 30] | 23.5 [18 to 34] | 18 [15 to 24] | 16.5 [13.5 to 27.5]
  AST (U/L)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  AST (U/L)- Day 308 | 17 [16 to 19] | 21 [18 to 27] | 18 [18 to 26] | 18 [14.5 to 21]
  Alkaline Phosphatase (U/L)- Screening | 57.5 [48.5 to 89.5] | 61 [53 to 74] | 64 [54.5 to 76] | 79 [64 to 81]
  Alkaline Phosphatase (U/L)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  Alkaline Phosphatase (U/L)- Day 14 | 53.5 [44 to 83.5] | 60 [53 to 69.5] | 62 [51 to 79] | 76 [59 to 77]
  Alkaline Phosphatase (U/L)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  Alkaline Phosphatase (U/L)- Day 70 | 63 [42 to 82] | 62 [49 to 70] | 63 [52 to 77] | 60.5 [44 to 74.5]
  Alkaline Phosphatase (U/L)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  Alkaline Phosphatase (U/L)- Day 126 | 59 [46 to 85] | 60.5 [52 to 77] | 64 [53 to 79] | 64 [50 to 73]
  Alkaline Phosphatase (U/L)- Day 238: number analyzed (Participants) | 17 | 18 | 18 | 4
  Alkaline Phosphatase (U/L)- Day 238 | 65 [44 to 78] | 58 [52 to 66] | 67.5 [46 to 76] | 59 [48.5 to 80]
  Alkaline Phosphatase (U/L)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  Alkaline Phosphatase (U/L)- Day 308 | 60 [40 to 77] | 59 [51.5 to 70] | 60 [52 to 77] | 66.5 [51 to 87]

17. Primary Outcome: Part B Chemistry and Hematology Laboratory Measures, for Each Boost: Hemoglobin, Creatinine in g/dL
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, 8, and at Month 11
Population: T5-T8 All enrolled
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
g/dL
  Hemoglobin (g/dL)- Screening | 13.7 [13.25 to 15.05] | 14.65 [13.7 to 15.25] | 14.35 [13.05 to 15.05] | 14.2 [13.3 to 15.3]
  Hemoglobin (g/dL)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  Hemoglobin (g/dL)- Day 14 | 13.7 [12.9 to 14.5] | 14.05 [13.1 to 14.95] | 13.4 [12.1 to 14.5] | 13.8 [13.6 to 14.6]
  Hemoglobin (g/dL)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  Hemoglobin (g/dL)- Day 70 | 13.9 [13.2 to 14.8] | 13.9 [12.5 to 15.2] | 14 [12.1 to 15] | 13.65 [11.55 to 14.7]
  Hemoglobin (g/dL)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  Hemoglobin (g/dL)- Day 126 | 14 [13.4 to 15] | 14.45 [13 to 15.5] | 13.9 [13.2 to 14.5] | 13.75 [12.55 to 14.95]
  Hemoglobin (g/dL)- Day 238: number analyzed (Participants) | 18 | 18 | 18 | 4
  Hemoglobin (g/dL)- Day 238 | 13.55 [12.8 to 13.9] | 14.1 [12.1 to 14.9] | 13.8 [12.4 to 14.5] | 13.8 [12.1 to 15.05]
  Hemoglobin (g/dL)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  Hemoglobin (g/dL)- Day 308 | 13.45 [12.6 to 14.6] | 14.55 [13.1 to 15.3] | 14.1 [12.7 to 14.6] | 14.1 [12.8 to 15.05]
  Creatinine (g/dL)- Screening | 0.00086 [0.00075 to 0.00093] | 0.00088 [0.00079 to 0.00094] | 0.00087 [0.000775 to 0.000985] | 0.00081 [0.0007 to 0.00084]
  Creatinine (g/dL)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  Creatinine (g/dL)- Day 14 | 0.00093 [0.00077 to 0.00101] | 0.000875 [0.00077 to 0.000945] | 0.00085 [0.0008 to 0.00101] | 0.00095 [0.00073 to 0.00098]
  Creatinine (g/dL)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  Creatinine (g/dL)- Day 70 | 0.00089 [0.00082 to 0.00103] | 0.0009 [0.00074 to 0.00095] | 0.0009 [0.00082 to 0.00102] | 0.000765 [0.00068 to 0.0009]
  Creatinine (g/dL)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  Creatinine (g/dL)- Day 126 | 0.0009 [0.00072 to 0.001] | 0.000895 [0.00079 to 0.001005] | 0.00093 [0.00081 to 0.00098] | 0.000765 [0.00064 to 0.000995]
  Creatinine (g/dL)- Day 238: number analyzed (Participants) | 17 | 18 | 18 | 4
  Creatinine (g/dL)- Day 238 | 0.0009 [0.00076 to 0.00101] | 0.000885 [0.00076 to 0.00098] | 0.00087 [0.0008 to 0.00097] | 0.00082 [0.0007 to 0.000955]
  Creatinine (g/dL)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  Creatinine (g/dL)- Day 308 | 0.0009 [0.00073 to 0.00101] | 0.00082 [0.00079 to 0.001015] | 0.0009 [0.0008 to 0.00096] | 0.00087 [0.00073 to 0.000995]

18. Primary Outcome: Part B Chemistry and Hematology Laboratory Measures
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, 8, and at Month 11
Population: T5-T8 All enrolled
Measure: Median (Inter-Quartile Range); unit: 1000 cells per mm^3
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
1000 cells per mm^3
  WBC (1000 cells per mm^3)- Screening | 5.63 [4.66 to 7.05] | 6.15 [5.15 to 7.1] | 6.12 [5.1 to 7.55] | 6.9 [6.17 to 8]
  WBC (1000 cells per mm^3)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  WBC (1000 cells per mm^3)- Day 14 | 5.695 [4.825 to 7.49] | 5.95 [4.75 to 6.75] | 6.1 [4.9 to 7.17] | 5.27 [5.04 to 5.8]
  WBC (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  WBC (1000 cells per mm^3)- Day 70 | 5.5 [4.9 to 7.46] | 5.7 [5.1 to 7.5] | 6 [5.3 to 7.62] | 5.13 [4.43 to 5.9]
  WBC (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  WBC (1000 cells per mm^3)- Day 126 | 6 [4.53 to 6.74] | 6.33 [5.55 to 8] | 6.67 [5.35 to 7.06] | 5.49 [4.8 to 6.34]
  WBC (1000 cells per mm^3)- Day 238: number analyzed (Participants) | 18 | 18 | 18 | 4
  WBC (1000 cells per mm^3)- Day 238 | 5.935 [4.8 to 7.38] | 5.75 [4.69 to 6.5] | 5.98 [5.3 to 6.5] | 5.615 [5.1 to 6.715]
  WBC (1000 cells per mm^3)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  WBC (1000 cells per mm^3)- Day 308 | 5.39 [4.7 to 7.06] | 5.95 [5.11 to 6.845] | 5.6 [5.12 to 7.19] | 7.33 [5.8 to 8.68]
  Neutrophils (1000 cells per mm^3)- Screening | 3.0445 [2.7 to 4.272] | 3.718 [2.676 to 4.5425] | 3.805 [2.946 to 4.803] | 4.361 [3.625 to 5.232]
  Neutrophils (1000 cells per mm^3)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  Neutrophils (1000 cells per mm^3)- Day 14 | 3.1395 [2.455 to 4.45] | 3.375 [2.255 to 4.1685] | 3.44 [2.72 to 4.55] | 3.029 [2.53 to 3.631]
  Neutrophils (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  Neutrophils (1000 cells per mm^3)- Day 70 | 2.97 [2.48 to 4.25] | 3.09 [2.46 to 4.8] | 3.49 [3.02 to 5.039] | 2.9985 [2.6275 to 3.265]
  Neutrophils (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  Neutrophils (1000 cells per mm^3)- Day 126 | 2.76 [2.49 to 4.11] | 3.61 [3.006 to 4.9155] | 3.7 [3.375 to 4.32] | 3.3835 [2.9735 to 3.867]
  Neutrophils (1000 cells per mm^3)- Day 238: number analyzed (Participants) | 17 | 18 | 18 | 4
  Neutrophils (1000 cells per mm^3)- Day 238 | 3.16 [2.29 to 4.25] | 3.2765 [2.537 to 4.019] | 3.245 [2.9 to 4.1] | 3.0805 [2.9585 to 3.9365]
  Neutrophils (1000 cells per mm^3)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  Neutrophils (1000 cells per mm^3)- Day 308 | 3.133 [2.24 to 3.48] | 3.663 [2.655 to 4.341] | 3.416 [2.81 to 4.488] | 4.225 [3.5265 to 5.681]
  Lymphocytes (1000 cells per mm^3)- Screening | 1.805 [1.72 to 2.145] | 2.0365 [1.575 to 2.1045] | 1.8095 [1.463 to 2.245] | 1.918 [1.42 to 2.072]
  Lymphocytes (1000 cells per mm^3)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  Lymphocytes (1000 cells per mm^3)- Day 14 | 1.9705 [1.585 to 2.2425] | 1.94 [1.6 to 2.11] | 1.89 [1.458 to 2.13] | 1.72 [1.618 to 1.936]
  Lymphocytes (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  Lymphocytes (1000 cells per mm^3)- Day 70 | 1.99 [1.54 to 2.37] | 1.986 [1.68 to 2.32] | 1.76 [1.344 to 2.451] | 1.619 [1.1685 to 2.0525]
  Lymphocytes (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  Lymphocytes (1000 cells per mm^3)- Day 126 | 1.8 [1.58 to 2.33] | 2.025 [1.84 to 2.199] | 1.99 [1.265 to 2.36] | 1.553 [1.3175 to 1.729]
  Lymphocytes (1000 cells per mm^3)- Day 238: number analyzed (Participants) | 17 | 18 | 18 | 4
  Lymphocytes (1000 cells per mm^3)- Day 238 | 1.85 [1.6 to 2.04] | 1.78 [1.64 to 2.022] | 1.885 [1.65 to 2.242] | 1.836 [1.534 to 2.1425]
  Lymphocytes (1000 cells per mm^3)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  Lymphocytes (1000 cells per mm^3)- Day 308 | 1.805 [1.71 to 1.989] | 1.816 [1.4885 to 2.229] | 1.72 [1.377 to 2.06] | 2.0175 [1.6075 to 2.2275]
  Platelets (1000 cells per mm^3)- Screening | 246.5 [214.5 to 268.5] | 284.5 [240.5 to 314] | 274 [237 to 327] | 269 [223.6 to 280]
  Platelets (1000 cells per mm^3)- Day 14: number analyzed (Participants) | 20 | 20 | 19 | 5
  Platelets (1000 cells per mm^3)- Day 14 | 258.5 [213.5 to 285.5] | 269 [240 to 300.5] | 274 [242.5 to 320] | 281 [277 to 297.1]
  Platelets (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 19 | 19 | 19 | 4
  Platelets (1000 cells per mm^3)- Day 70 | 253 [217 to 269] | 272 [213 to 308] | 277.3 [244 to 311] | 229.05 [189.55 to 272]
  Platelets (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 19 | 20 | 19 | 4
  Platelets (1000 cells per mm^3)- Day 126 | 241 [219 to 298] | 286.5 [236.5 to 310] | 265 [247 to 346] | 244.85 [193.85 to 287.5]
  Platelets (1000 cells per mm^3)- Day 238: number analyzed (Participants) | 18 | 18 | 18 | 4
  Platelets (1000 cells per mm^3)- Day 238 | 248 [227 to 270] | 262.5 [232 to 298] | 272.3 [258 to 332] | 242.3 [208.3 to 313.5]
  Platelets (1000 cells per mm^3)- Day 308: number analyzed (Participants) | 18 | 20 | 19 | 4
  Platelets (1000 cells per mm^3)- Day 308 | 229.5 [211 to 264] | 282 [217.5 to 306.5] | 274.9 [228 to 303] | 262.9 [202.4 to 297]

19. Primary Outcome: Part B Magnitude and Breadth of Neutralizing Antibody Response Against Autologous Viral Isolates and Related CH103 and CH235 Precursor Detection Isolates 2 Weeks After the Fourth Vaccinations
Description: Magnitude-breadth characterize the magnitude (ID50) and breadth (number of virus isolates) of each individual serum sample assayed against a panel of virus isolates. MB curves show, for each possible magnitude threshold, the proportion of isolates among the virus panel with magnitudes greater than this threshold. The area under the magnitude-breadth curve (AUC-MB) integrates magnitude and breadth information and provides effective tools to display, summarize, and compare multi-viral immunological data in the context of HIV-1 vaccine trials.
Time Frame: Measured at Month 8.5
Measure: Median (Inter-Quartile Range); unit: log10 titer*percentage of isolates
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
log10 titer*percentage of isolates | 1.1384246921 [1.0811824148 to 1.1585691555] | 1.1849438379 [1.1769724686 to 1.219004435] | 1.1194766117 [1.050817124 to 1.1611045902] | 0.6989700043 [0.6989700043 to 0.6989700043]

20. Primary Outcome: Part B Magnitude and Breadth of Neutralizing Antibody Responses Against a Panel of Heterologous Tier 2 Isolates Induced 2 Weeks After the Fourth Vaccinations
Description: as for outcome 19
Time Frame: Measured at Month 8.5
Measure: Median (Inter-Quartile Range); unit: log10 titer*percentage of isolates
Arm/Group | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 5
log10 titer*percentage of isolates | 0.6989700043 [0.6989700043 to 0.6989700043] | 0.7500872649 [0.6989700043 to 0.8869830068] | 0.6989700043 [0.6989700043 to 0.7983235391] | 0.6989700043 [0.6989700043 to 0.7487297683]

21. Primary Outcome: Number of Part C Participants Reporting Local Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through Month Measured through Month Measured through 7 days after the vaccination at Month 0, 2, 4
Measure: Count of Participants; unit: Participants
Groups:
- Group 9: Vaccine: 400mcg CH505TF(m0), 400mcg CH505w53(m2), 400mcg CH505w78(m4)
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
Participants
  Pain: None | 1
  Pain: Mild | 6
  Pain: Moderate | 3
  Pain: Severe | 0
  Pain: Potentially Life-threatening | 0
  Tenderness: None | 1
  Tenderness: Mild | 6
  Tenderness: Moderate | 3
  Tenderness: Severe | 0
  Tenderness: Potentially Life-threatening | 0
  Pain and/or Tenderness: None | 1
  Pain and/or Tenderness: Mild | 5
  Pain and/or Tenderness: Moderate | 4
  Pain and/or Tenderness: Severe | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0
  Erythema/Redness: None | 7
  Erythema/Redness: Mild | 1
  Erythema/Redness: Moderate | 2
  Erythema/Redness: Severe | 0
  Erythema/Redness: Potentially Life-threatening | 0
  Induration/Swelling: None | 5
  Induration/Swelling: Mild | 2
  Induration/Swelling: Moderate | 3
  Induration/Swelling: Severe | 0
  Induration/Swelling: Potentially Life-threatening | 0
  Erythema and/or Induration: None | 5
  Erythema and/or Induration: Mild | 2
  Erythema and/or Induration: Moderate | 3
  Erythema and/or Induration: Severe | 0
  Erythema and/or Induration: Potentially Life-threatening | 0

22. Primary Outcome: Number of Part C Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through Month Measured through Month Measured through 7 days after the vaccination at Month 0, 2, 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
Participants
  Malaise and/or fatigue: None | 2
  Malaise and/or fatigue: Mild | 4
  Malaise and/or fatigue: Moderate | 4
  Malaise and/or fatigue: Severe | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0
  Myalgia: None | 5
  Myalgia: Mild | 3
  Myalgia: Moderate | 2
  Myalgia: Severe | 0
  Myalgia: Potentially Life-threatening | 0
  Headache: None | 4
  Headache: Mild | 5
  Headache: Moderate | 1
  Headache: Severe | 0
  Headache: Potentially Life-threatening | 0
  Nausea: None | 4
  Nausea: Mild | 4
  Nausea: Moderate | 2
  Nausea: Severe | 0
  Nausea: Potentially Life-threatening | 0
  Vomiting: None | 10
  Vomiting: Mild | 0
  Vomiting: Moderate | 0
  Vomiting: Severe | 0
  Vomiting: Potentially Life-threatening | 0
  Chills: None | 9
  Chills: Mild | 1
  Chills: Moderate | 0
  Chills: Severe | 0
  Chills: Potentially Life-threatening | 0
  Arthralgia: None | 7
  Arthralgia: Mild | 0
  Arthralgia: Moderate | 3
  Arthralgia: Severe | 0
  Arthralgia: Potentially Life-threatening | 0
  Max. Systemic Symptoms: None | 2
  Max. Systemic Symptoms: Mild | 4
  Max. Systemic Symptoms: Moderate | 4
  Max. Systemic Symptoms: Severe | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0
  Temperature: None | 9
  Temperature: Mild | 1
  Temperature: Moderate | 0
  Temperature: Severe | 0
  Temperature: Potentially Life-threatening | 0

23. Primary Outcome: Part C: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity During the Vaccine Regime
Description: as for outcome 3
Time Frame: Measured through Month 16
Measure: Count of Participants; unit: Participants
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
Participants | 0

24. Primary Outcome: Number of Part C Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through the Month 4 administration
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
Participants
  Reactogenicity symptoms | 0
  Withdrawal by Subject | 1
  Investigator reason | 0
  Lost to Follow-Up | 0
  Did not discontinue SPA | 9

25. Primary Outcome: Part C Chemistry and Hematology Laboratory Measures, for Each Boost: Alkaline Phosphatase, AST, ALT in U/L
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, and at Month 10
Population: T9 All enrolled
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
U/L
  ALT (SGPT) (U/L)- Screening | 13 [12 to 15]
  ALT (SGPT) (U/L)- Day 14 | 13 [12 to 15]
  ALT (SGPT) (U/L)- Day 70: number analyzed (Participants) | 9
  ALT (SGPT) (U/L)- Day 70 | 14 [13 to 14]
  ALT (SGPT) (U/L)- Day 126: number analyzed (Participants) | 9
  ALT (SGPT) (U/L)- Day 126 | 13 [11 to 15]
  ALT (SGPT) (U/L)- Day 303: number analyzed (Participants) | 9
  ALT (SGPT) (U/L)- Day 303 | 14 [11 to 15]
  AST (U/L)- Screening | 17.5 [16 to 21]
  AST (U/L)- Day 14 | 16 [14 to 18]
  AST (U/L)- Day 70: number analyzed (Participants) | 9
  AST (U/L)- Day 70 | 16 [15 to 20]
  AST (U/L)- Day 126: number analyzed (Participants) | 9
  AST (U/L)- Day 126 | 14 [13 to 16]
  AST (U/L)- Day 303: number analyzed (Participants) | 9
  AST (U/L)- Day 303 | 16 [15 to 17]
  Alkaline Phosphatase (U/L)- Screening | 73.5 [50 to 85]
  Alkaline Phosphatase (U/L)- Day 14 | 60 [54 to 66]
  Alkaline Phosphatase (U/L)- Day 70: number analyzed (Participants) | 9
  Alkaline Phosphatase (U/L)- Day 70 | 63 [57 to 72]
  Alkaline Phosphatase (U/L)- Day 126: number analyzed (Participants) | 9
  Alkaline Phosphatase (U/L)- Day 126 | 61 [56 to 76]
  Alkaline Phosphatase (U/L)- Day 303: number analyzed (Participants) | 9
  Alkaline Phosphatase (U/L)- Day 303 | 63 [53 to 71]

26. Primary Outcome: Part C Chemistry and Hematology Laboratory Measures, for Each Boost: Hemoglobin, Creatinine in g/dL
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, and at Month 10
Population: T9 All enrolled
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
g/dL
  Hemoglobin (g/dL)- Screening | 14.45 [13.3 to 15.1]
  Hemoglobin (g/dL)- Day 14 | 13.85 [13 to 15.1]
  Hemoglobin (g/dL)- Day 70: number analyzed (Participants) | 9
  Hemoglobin (g/dL)- Day 70 | 14.3 [13.6 to 14.6]
  Hemoglobin (g/dL)- Day 126: number analyzed (Participants) | 9
  Hemoglobin (g/dL)- Day 126 | 13.9 [13.2 to 14.2]
  Hemoglobin (g/dL)- Day 303: number analyzed (Participants) | 9
  Hemoglobin (g/dL)- Day 303 | 13.6 [13.2 to 14.6]
  Creatinine (g/dL)- Screening | 0.000815 [0.00078 to 0.00089]
  Creatinine (g/dL)- Day 14 | 0.00082 [0.00077 to 0.00088]
  Creatinine (g/dL)- Day 70: number analyzed (Participants) | 9
  Creatinine (g/dL)- Day 70 | 0.0008 [0.00076 to 0.0009]
  Creatinine (g/dL)- Day 126: number analyzed (Participants) | 9
  Creatinine (g/dL)- Day 126 | 0.00083 [0.00077 to 0.00091]
  Creatinine (g/dL)- Day 303: number analyzed (Participants) | 9
  Creatinine (g/dL)- Day 303 | 0.00084 [0.00074 to 0.00089]

27. Primary Outcome: Part C Chemistry and Hematology Laboratory Measures
Description: as for outcome 5
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 2, 4, and at Month 10
Population: T9 All enrolled
Measure: Median (Inter-Quartile Range); unit: 1000 cells per mm^3
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
1000 cells per mm^3
  WBC (1000 cells per mm^3)- Screening | 5.95 [4.94 to 8.03]
  WBC (1000 cells per mm^3)- Day 14 | 6.08 [4.56 to 7.2]
  WBC (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 9
  WBC (1000 cells per mm^3)- Day 70 | 6.67 [4.53 to 9.08]
  WBC (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 9
  WBC (1000 cells per mm^3)- Day 126 | 6.2 [4.31 to 7.17]
  WBC (1000 cells per mm^3)- Day 303: number analyzed (Participants) | 9
  WBC (1000 cells per mm^3)- Day 303 | 7.62 [4.36 to 8.4]
  Neutrophils (1000 cells per mm^3)- Screening | 3.783 [2.97 to 4.79]
  Neutrophils (1000 cells per mm^3)- Day 14 | 3.47 [2.83 to 4.33]
  Neutrophils (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 9
  Neutrophils (1000 cells per mm^3)- Day 70 | 3.5 [2.71 to 5.88]
  Neutrophils (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 9
  Neutrophils (1000 cells per mm^3)- Day 126 | 3.639 [2.55 to 3.98]
  Neutrophils (1000 cells per mm^3)- Day 303: number analyzed (Participants) | 9
  Neutrophils (1000 cells per mm^3)- Day 303 | 4.58 [2.53 to 5.8]
  Lymphocytes (1000 cells per mm^3)- Screening | 1.6835 [1.4 to 2.4]
  Lymphocytes (1000 cells per mm^3)- Day 14 | 1.629 [1.25 to 2.11]
  Lymphocytes (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 9
  Lymphocytes (1000 cells per mm^3)- Day 70 | 1.73 [1.28 to 2.33]
  Lymphocytes (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 9
  Lymphocytes (1000 cells per mm^3)- Day 126 | 1.562 [1.41 to 2.2]
  Lymphocytes (1000 cells per mm^3)- Day 303: number analyzed (Participants) | 9
  Lymphocytes (1000 cells per mm^3)- Day 303 | 1.806 [1.295 to 2.1]
  Platelets (1000 cells per mm^3)- Screening | 276.5 [220 to 334]
  Platelets (1000 cells per mm^3)- Day 14 | 299 [240 to 320]
  Platelets (1000 cells per mm^3)- Day 70: number analyzed (Participants) | 9
  Platelets (1000 cells per mm^3)- Day 70 | 288 [260 to 319]
  Platelets (1000 cells per mm^3)- Day 126: number analyzed (Participants) | 9
  Platelets (1000 cells per mm^3)- Day 126 | 275 [233 to 316]
  Platelets (1000 cells per mm^3)- Day 303: number analyzed (Participants) | 9
  Platelets (1000 cells per mm^3)- Day 303 | 280 [233 to 295]

28. Secondary Outcome: Part C Magnitude and Breadth of Neutralizing Antibody Response Against Autologous Viral Isolates and Related CH103 and CH235 Precursor Detection Isolates 2 Weeks After the Third (Final) Vaccination
Description: Magnitude-breadth characterize the magnitude (ID50) and breadth (number of virus isolates) of each individual serum sample assayed against a panel of virus isolates. MB curves show, for each possible magnitude threshold, the proportion of isolates among the virus panel with magnitudes greater than this threshold. The area under the magnitude-breadth curve (AUC-MB) integrates magnitude and breadth information and provides effective tools to display, summarize, and compare multi-viral immunological data in the context of HIV-1 vaccine trials. Six autologous isolates were assayed and included for the AUC-MB calculation: CH0505.w4.3, CH0505.w53.16, CH0505.w78.e33, CH0505.w100.B6, CH0505s, and CH0505TF.M5.
Time Frame: Measured at Month 4.5
Measure: Median (Inter-Quartile Range); unit: log10 titer*percentage of isolates
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
log10 titer*percentage of isolates | 0.9919921716 [0.9551699712 to 1.0164352642]

29. Secondary Outcome: Part C Magnitude and Breadth of Neutralizing Antibody Responses Against a Panel of Heterologous Tier 2 Isolates Induced 2 Weeks After the Third (Final) Vaccination
Description: as for outcome 28
Time Frame: Measured at Month 4.5
Measure: Median (Inter-Quartile Range); unit: log10 titer*percentage of isolates
Arm/Group | Group 9: Vaccine
Number analyzed (Participants) | 10
log10 titer*percentage of isolates | 0.8284675826 [0.6989700043 to 0.8446388582]

30. Secondary Outcome: Part A: Occurence of Memory B Cells Differentially Binding to the CH505 Wildtype gp120 TF Env vs the Mutant CH505 Env I Delta 371 gp120 2 Weeks After the Third Vaccination With CH505TF gp120
Description: The CD4 binding-site (CD4bs) and Env-specific B cells were quantified using biotinylated CH505TF gp120 protein probes and the CD4bs-mutant in the context of a flow cytometry panel to identify and characterize those B cells. Post-vaccine samples are defined as positive responders if the frequency of Env-specific B cells for the post-vaccine data was statistically greater than that for the data from baseline, compared by one-sided Fisher's exact test. The Fisher's exact test is not applied to compare between endpoints.
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  CD4bs+ CH505+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CD4bs+ CH505+ B cells | 9 | 9 | 11 | 0
  CD4bs+ CH505+ IgG+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CD4bs+ CH505+ IgG+ B cells | 10 | 9 | 11 | 0
  CH505+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH505+ B cells | 11 | 11 | 12 | 0
  CH505+ IgG+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH505+ IgG+ B cells | 11 | 11 | 12 | 0

31. Secondary Outcome: Part A: Level of Memory B Cells Differentially Binding to the CH505 Wildtype gp120 TF Env vs the Mutant CH505 Env I Delta 371 gp120 2 Weeks After the Third Vaccination With CH505TF gp120
Description: The CD4 binding-site (CD4bs) and Env-specific B cells were quantified using biotinylated CH505TF gp120 protein probes and the CD4bs-mutant in the context of a flow cytometry panel to identify and characterize those B cells. The reported frequencies are: The % CH505+ of total B cells equals the frequency of double-positive CH505 gp120+ B cells out of total B cells; the % CD4bs CH505+ of total B cells equals the frequency of double-positive CH505 gp120+ B cells that are negative for the CD4bs mutant (CH505 I delta 371) out of total B cells; the % CH505+ of IgG+ B cells equals the frequency of double-positive CH505 gp120+ IgG+ B cells out of IgG+ B cells; and the % CD4bs CH505+ of IgG+ B cells equals the frequency of double-positive CH505 gp120+ IgG+ B cells that are negative for the CD4bs mutant (CH505 I delta 371) out of IgG+ B cells.
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: % B-cells
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
% B-cells
  CD4bs+ CH505+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CD4bs+ CH505+ B cells | 0.0336336336 [0.015625 to 0.0450757377] | 0.0383802953 [0.0260133882 to 0.0607006346] | 0.033951166 [0.0243709361 to 0.0960959665] | 0.0052190432 [0.001061008 to 0.0127753304]
  CD4bs+ CH505+ IgG+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CD4bs+ CH505+ IgG+ B cells | 0.3432494279 [0.0737350136 to 0.6560563723] | 0.2227163176 [0.0869480928 to 0.3467235194] | 0.2295544376 [0.1114627336 to 0.5010063155] | 0.001277025 [0 to 0.0061192021]
  CH505+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH505+ B cells | 0.3928819444 [0.248440694 to 0.7179063361] | 0.5019394658 [0.186793809 to 0.895629002] | 0.6492676935 [0.3473426094 to 1.1017202497] | 0.0062628519 [0.0018567639 to 0.013876652]
  CH505+ IgG+ B cells: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH505+ IgG+ B cells | 3.9065053939 [2.8087107152 to 5.6719558166] | 3.4168305845 [1.2972281912 to 5.4550889701] | 4.0027261874 [3.0877152432 to 6.7554425115] | 0.0051081002 [0 to 0.0122384041]

32. Secondary Outcome: Part A: Magnitude and Breadth of Neutralizing Antibody Responses Against Autologous Viral Isolates as Assessed by Area Under the Magnitude-breadth Curves 2 Weeks After the Third Vaccination With CH505TF gp120
Description: as for outcome 28
Time Frame: Measured at Month 4.5
Population: Only participants with data available for all six isolates are included.
Measure: Mean (Inter-Quartile Range); unit: log10 titer*percentage of isolates
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
log10 titer*percentage of isolates | 0.94 [0.88 to 0.97] | 0.93 [0.85 to 0.97] | 0.97 [0.95 to 1.01] | 0.70 [0.70 to 0.70]

33. Secondary Outcome: Part A: Occurrence of CD4+ T-cell Responses as Assessed by Intracellular Cytokine Staining Assays (ICS) 2 Weeks After the Third and Fifth Vaccination With CH505TF
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. Response positivity is derived by testing if the number of cells expressing the marker is equal in the stimulated vs. unstimulated cells. Response is positive if the one-sided Fisher's exact test (discrete Bonferroni adjustment over the peptide pools) p greater than or equal to 0.00001. The Fisher's exact test is not applied to compare between endpoints. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high.
Time Frame: Measured at Months 4.5 and 12.5
Population: "Overall Number of Participants Analyzed" includes the HIV uninfected participants with samples collected at the months 4.5 and 12.5 immunogenicity timepoint. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  Any Env at Month 4.5: number analyzed (Participants) | 11 | 10 | 12 | 3
  Any Env at Month 4.5 | 4 | 6 | 5 | 0
  Any Env at Month 12.5: number analyzed (Participants) | 9 | 9 | 11 | 3
  Any Env at Month 12.5 | 4 | 2 | 0 | 0
  Env-1-PTEg-SEQ at Month 4.5: number analyzed (Participants) | 11 | 10 | 12 | 3
  Env-1-PTEg-SEQ at Month 4.5 | 4 | 6 | 5 | 0
  Env-1-PTEg-SEQ at Month 12.5: number analyzed (Participants) | 9 | 9 | 11 | 3
  Env-1-PTEg-SEQ at Month 12.5 | 4 | 2 | 0 | 0
  Env-2-PTEg-SEQ at Month 4.5: number analyzed (Participants) | 11 | 10 | 12 | 3
  Env-2-PTEg-SEQ at Month 4.5 | 1 | 6 | 3 | 0
  Env-2-PTEg-SEQ at Month 12.5: number analyzed (Participants) | 9 | 9 | 11 | 3
  Env-2-PTEg-SEQ at Month 12.5 | 2 | 2 | 0 | 0

34. Secondary Outcome: Part A: Level of CD4+ T-cell Responses as Assessed by Intracellular Cytokine Staining Assays (ICS) 2 Weeks After the Third and Fifth Vaccination With CH505TF
Description: as for outcome 33
Time Frame: Measured at Months 4.5 and 12.5
Population: as for outcome 33
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
% CD4+ T-cells
  Any Env at Month 4.5: number analyzed (Participants) | 11 | 10 | 12 | 3
  Any Env at Month 4.5 | 0.07193596 [0.0453187 to 0.11852354] | 0.132646355 [0.04007281 to 0.37230634] | 0.073603225 [0.031028225 to 0.158387505] | 0.00911761 [-0.00401237 to 0.02455366]
  Any Env at Month 12.5: number analyzed (Participants) | 9 | 9 | 11 | 3
  Any Env at Month 12.5 | 0.07052576 [0.05099588 to 0.08964846] | 0.04367241 [0.04052204 to 0.07384431] | 0.04605537 [0.02988448 to 0.07826411] | -0.00279413 [-0.00571998 to 0.01167789]
  Env-1-PTEg-SEQ at Month 4.5: number analyzed (Participants) | 11 | 10 | 12 | 3
  Env-1-PTEg-SEQ at Month 4.5 | 0.04602687 [0.02316902 to 0.08966309] | 0.0783176 [0.02824605 to 0.1525245] | 0.04050064 [0.014047985 to 0.105562815] | -0.00285989 [-0.0052998 to 0.0234871]
  Env-1-PTEg-SEQ at Month 12.5: number analyzed (Participants) | 9 | 9 | 11 | 3
  Env-1-PTEg-SEQ at Month 12.5 | 0.04420066 [0.03908209 to 0.06830406] | 0.02299821 [0.01601415 to 0.0551526] | 0.02889892 [0.00559549 to 0.05235601] | 0.00867745 [0.00277486 to 0.0127573]
  Env-2-PTEg-SEQ at Month 4.5: number analyzed (Participants) | 11 | 10 | 12 | 3
  Env-2-PTEg-SEQ at Month 4.5 | 0.02507079 [0.01127097 to 0.03920034] | 0.048858555 [0.01152919 to 0.13757644] | 0.021711805 [0.00698941 to 0.06117293] | 0.00128743 [0.00106656 to 0.0119775]
  Env-2-PTEg-SEQ at Month 12.5: number analyzed (Participants) | 9 | 9 | 11 | 3
  Env-2-PTEg-SEQ at Month 12.5 | 0.0213444 [0.00876609 to 0.06531986] | 0.02479532 [0.01261996 to 0.02788738] | 0.02428899 [0.0057976 to 0.04546687] | -0.00849484 [-0.01147158 to -0.00107941]

35. Secondary Outcome: Part A: Occurrence of Monoclonal Antibodies Evaluated for CD4 Binding Site Loop Binding
Description: ELISA responses were measured at serial three-fold serum dilutions from 1:30 to 1:(30×3^11 = 5,314,410) for each analyte. Positive responses are defined as (analyte OD) > 3×(background OD) in wells of dilutions 1:30 and 1:90.
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Participants
  CH0505_CON D7 gp120_avi/293F/Mon: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH0505_CON D7 gp120_avi/293F/Mon | 11 | 11 | 12 | 0
  CH0505_CON D7gp120_D368R_avi/293F/Mon: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH0505_CON D7gp120_D368R_avi/293F/Mon | 11 | 11 | 12 | 0
  CH505TF_D7gp120d371_avi: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH505TF_D7gp120d371_avi | 11 | 11 | 12 | 0

36. Secondary Outcome: Part A: Level of Monoclonal Antibodies Evaluated for CD4 Binding Site Loop Binding
Description: ELISA responses were measured at serial three-fold serum dilutions from 1:30 to 1:(30×3^11 = 5,314,410) for each analyte. The area under the dilution-magnitude curve (AUC) was calculated as the average untransformed optical density (OD) over the log10 dilutions using the trapezoidal rule.
Time Frame: Measured at Month 4.5
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Optical density
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Vaccine | Part A, Group 4: Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 6
Optical density
  CH0505_CON D7 gp120_avi/293F/Mon: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH0505_CON D7 gp120_avi/293F/Mon | 6.6971124919 [5.4824094895 to 7.4119832678] | 6.8592025102 [5.1850198115 to 7.5037456131] | 7.5422612265 [7.2787233014 to 8.1849197005] | 0.229304475 [0.225129664 to 0.3374678635]
  CH0505_CON D7gp120_D368R_avi/293F/Mon: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH0505_CON D7gp120_D368R_avi/293F/Mon | 6.1512380643 [5.2453995062 to 7.2585410723] | 6.5292373784 [4.7412493324 to 7.2369990477] | 7.3797656551 [6.9723160316 to 7.907127778] | 0.2318809298 [0.230807407 to 0.3256591124]
  CH505TF_D7gp120d371_avi: number analyzed (Participants) | 11 | 12 | 12 | 3
  CH505TF_D7gp120d371_avi | 5.6756913098 [4.905379044 to 7.1963244607] | 6.1353499266 [4.3269053068 to 6.8560177258] | 6.7855111323 [6.4254992896 to 7.2542946932] | 0.2366759984 [0.2306881267 to 0.3305018931]

37. Secondary Outcome: Part B: HIV-specific Binding Ab Responses as Assessed by Binding Ab Multiplex Assay 2 Weeks After the Second and After the Fourth Vaccinations
Description: as for outcome 10
Time Frame: Measured at Month 2.5 and Month 8.5
Reporting Status: Not Posted, anticipated posting 2024-07

38. Secondary Outcome: Part B: Occurrence of CD4+ T-cell Responses as Assessed by Intracellular Cytokine Staining (ICS) Assays 2 Weeks After the Second and Fourth (Final) Vaccinations With EnvSeq-1 Immunogens or CH505 M5 gp120
Description: as for outcome 33
Time Frame: Measured at Months 2.5 and 8.5
Reporting Status: Not Posted, anticipated posting 2024-07

39. Secondary Outcome: Part B: Level of CD4+ T-cell Responses as Assessed by Intracellular Cytokine Staining (ICS) Assays 2 Weeks After the Second and Fourth (Final) Vaccinations With EnvSeq-1 Immunogens or CH505 M5 gp120
Description: as for outcome 33
Time Frame: Measured at Months 2.5 and 8.5
Reporting Status: Not Posted, anticipated posting 2024-07

40. Secondary Outcome: Part B: Occurrence of Monoclonal Antibodies Evaluated for CD4 Binding Site Loop Binding
Description: as for outcome 35
Time Frame: Measured at Month 2.5
Reporting Status: Not Posted, anticipated posting 2024-07

41. Secondary Outcome: Part B: Level of Monoclonal Antibodies Evaluated for CD4 Binding Site Loop Binding
Description: as for outcome 36
Time Frame: Measured at Month 2.5
Reporting Status: Not Posted, anticipated posting 2024-07

42. Secondary Outcome: Part C: Percent B Cells Expressing Candidate CH103 Precursors With Immunogenetics, Function, and Structure Similar to CH103 Lineage Antibodies
Description: as for outcome 30
Time Frame: Measured at Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

43. Secondary Outcome: Part C: Alterations in Frequency of CH103-like Precursor B Cells Prior to CH505 TF (First) Vaccination and After the Final Vaccination
Description: as for outcome 30
Time Frame: Measured at Month 0 and at Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

44. Secondary Outcome: Part C: Characterization of B-cell Derived Antibodies (Binding, Neutralization and Structure Compared With the CH103 Lineage Members, Including the UCA)
Description: as for outcome 30
Time Frame: Measured at Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

45. Secondary Outcome: Part C: HIV-specific Binding Ab Responses as Assessed by Binding Ab Multiplex Assay 2 Weeks After the Final Vaccination
Description: as for outcome 8
Time Frame: Measured at Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

46. Secondary Outcome: Part C: Frequencies, Specificity and Phenotype of Vaccine-induced B-cell Responses as Measured by Multiparameter Flow Cytometry After Each Vaccination Compared to Baseline
Description: as for outcome 30
Time Frame: Measured at Month 0, Month 2.5 and Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

47. Secondary Outcome: Part C: Characterization of the B-cell Derived Antibodies (Binding of CH505 TF, wk53, wk78 Proteins), Neutralization of Autologous or Mutant CH505 Viruses, and Structure
Description: as for outcome 30
Time Frame: Measured at Month 0, Month 2.5 and Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

48. Secondary Outcome: Part C: Response Rate and Magnitude of CD4+ T-cell Responses as Assessed by ICS Assays 2 Weeks After the Final Vaccination
Description: as for outcome 33
Time Frame: Measured at Month 4.5
Reporting Status: Not Posted, anticipated posting 2024-07

ADVERSE EVENTS:
Time Frame: Serious Adverse events are collected throughout the study (months 0-18 for Part A, months 0-14 for Part B and months 0-10 for Part C). Non-serious adverse events are collected through 30 days after each vaccination (at months 0, 2, 4, 8, 12 for Part A, at months 0, 2, 4, 8 for Part B and months 0, 2, 4 for Part C).
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Placebo | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Group 8: Placebo | Group 9: Vaccine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/6 | 0/20 | 0/20 | 0/20 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12 | 0/6 | 1/20 | 0/20 | 0/20 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 4/12 | 8/12 | 7/12 | 4/6 | 15/20 | 17/20 | 18/20 | 3/5 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=12) | Group 2: Vaccine (N=12) | Group 3: Vaccine (N=12) | Group 4: Placebo (N=6) | Group 5: Vaccine (N=20) | Group 6: Vaccine (N=20) | Group 7: Vaccine (N=20) | Group 8: Placebo (N=5) | Group 9: Vaccine (N=10)
Any Event in SOC (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=12) | Group 2: Vaccine (N=12) | Group 3: Vaccine (N=12) | Group 4: Placebo (N=6) | Group 5: Vaccine (N=20) | Group 6: Vaccine (N=20) | Group 7: Vaccine (N=20) | Group 8: Placebo (N=5) | Group 9: Vaccine (N=10)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 6 (6) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 2 (5)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 2 (4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 3 (3) | 5 (8) | 3 (5) | 3 (6) | 12 (25) | 13 (21) | 9 (10) | 2 (2) | 6 (7)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 6 (6) | 3 (3) | 2 (2) | 3 (3)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Latent syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 1 (1) | 4 (8) | 1 (2) | 0 (0) | 3 (4) | 5 (8) | 3 (4) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Full blood count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Any Event in SOC (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Victim of sexual abuse (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03220724/Prot_SAP_ICF_000.pdf